CLINICAL TRIAL: NCT01281189
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of the Safety and Efficacy of Dexpramipexole in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Phase 3 Study of Dexpramipexole in ALS
Acronym: EMPOWER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 223AS302; EUDRA CT NO: 2010-022818-19
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Motor Neurone Disease; Motor Neuron Disease; Lou Gehrig's disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Dexpramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexpramipexole (Experimental)
  Interventions: Drug: Dexpramipexole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexpramipexole — Oral tablet 150mg twice daily for up to 18 months.
  Other Names: KNS-760704; BIIB050
  Arms: Dexpramipexole
Drug: Placebo — Oral tablet twice daily for up to 18 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether dexpramipexole (150 mg twice daily) is safe and effective in the treatment of Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a rapidly progressive, degenerative disease of motor neurons in the brain and spinal cord that leads to muscle atrophy and spasticity in limb and bulbar muscles resulting in weakness and loss of ambulation, oropharyngeal dysfunction, weight loss, and ultimately respiratory failure. The purpose of this study is to determine whether dexpramipexole (150 mg twice daily) is safe and effective in the treatment of ALS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years old, inclusive, on Day 1.
* Diagnosis of sporadic or familial ALS.
* Onset of first ALS symptoms within 24 months prior to Day 1.
* World Federation of Neurology El Escorial criteria are met for a possible, laboratory-supported probable, probable, or definite ALS diagnosis.
* Upright slow vital capacity (SVC) of 65% or more at screening.
* Patients taking or not taking Riluzole are eligible for this study: if a patient has never taken Riluzole, he or she is eligible; if a patient is currently taking Riluzole, he or she must have been on a stable dose for at least 60 days; if a patient has discontinued Riluzole, he or she must have stopped taking it for at least 30 days.
* Must be able to swallow tablets at the time of study entry.

Exclusion Criteria:

* Other medically significant illness.
* Clinically significant abnormal laboratory values.
* Pregnant women or women breastfeeding.
* Prior exposure to dexpramipexole.
* Currently taking pramipexole or other dopamine agonists.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 942 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, MSc, Principal Investigator — Professor of Neurology of the Harvard Medical School
Locations (82):
- United States (43):
  - Barrow Neurological Institute - St. Joseph's Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California at San Francisco - Fresno, Fresno, California
  - University of California, Irvine, Orange, California
  - University of California, Davis, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Hospital for Special Care, New Britain, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida Medical Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - St. Mary's Health Care, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Associates, P.C., Lincoln, Nebraska
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - Research Foundation of the State University of New York, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence ALS Center, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - ALS Center at Penn, Philadelphia, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Methodist Neurological Institute, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- Australia (4):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Calvary Health Care Bethlehem, Melbourne, Victoria
- Belgium (2):
  - AZ St-Lucas, Ghent
  - UZ Leuven, Leuven
- Canada (6):
  - Univ of Calgary / Foothills MC, Calgary, Alberta
  - CHUM - Hopital Notre Dame, Montreal, Quebec
  - Mcgill University, Montreal, Quebec
  - London Health Sciences Centre, London
  - Sunnybrook and Women's College and Health Sciences Centre, Toronto
  - University of British Columbia, Vancouver
- France (6):
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier La Timone, Marseille
  - CHU Gui de Chauliac, Montpellier
  - CHU de Nice - Hôpital de l'Archet 1, Nice
  - Hôpital La Pitié Salpétrière, Paris
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Bergmannsheil Gmbh, Bochum
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Jena, Jena
  - University of Ulm, RKU, Ulm
- Beaumont Hospital, Dublin, Ireland
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - UMC St. Radboud, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (4):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Carlos III, Madrid
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Solna, Stockholm
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Walton Centre for Neurology & Neurosurgery, Liverpool
  - Kings College Hospital NHS Foundation Trust, London
  - Newcastle University Hospital - Clinical Ageing Research Unit, Newcastle
  - John Radcliffe Hospital, Oxford
  - Sheffield Institute for Transnational Neuroscience, Sheffield

REFERENCES:
- [Derived] Cudkowicz ME, van den Berg LH, Shefner JM, Mitsumoto H, Mora JS, Ludolph A, Hardiman O, Bozik ME, Ingersoll EW, Archibald D, Meyers AL, Dong Y, Farwell WR, Kerr DA; EMPOWER investigators. Dexpramipexole versus placebo for patients with amyotrophic lateral sclerosis (EMPOWER): a randomised, double-blind, phase 3 trial. Lancet Neurol. 2013 Nov;12(11):1059-67. doi: 10.1016/S1474-4422(13)70221-7. Epub 2013 Sep 23. PMID 24067398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 942 participants (468 received placebo and 474 received dexpramipexole) recruited from 81 investigational sites in 11 countries worldwide. One additional participant was randomized in error and was not dosed. This subject was assigned to the placebo arm, but was removed from the intent-to-treat population as a result of the unintentional randomization performed in error by the site.
Groups:
- Placebo: Matching Placebo: Oral tablet twice daily.
- Dexpramipexole: Dexpramipexole: Oral tablet 150 mg twice daily. 300 mg/day
Period: Overall Study
Arm/Group | Placebo | Dexpramipexole
Started | 468 | 474
Completed | 321 | 331
Not Completed | 147 | 143
Not completed — Adverse Event | 7 | 9
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 21 | 24
Not completed — Physician Decision | 2 | 3
Not completed — Death | 103 | 91
Not completed — Other | 8 | 12

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population is defined as subjects who were randomized and received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexpramipexole | Total
Number analyzed (Participants) | 468 | 474 | 942
Age, Customized [Count of Participants; unit: Participants]
  Age (yrs): <50 | 114 | 114 | 228
  Age (yrs): 50-65 | 233 | 244 | 477
  Age (yrs): >65 | 121 | 116 | 237
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 167 | 337
  Male | 298 | 307 | 605
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 7 | 4 | 11
  Race: Black or African American | 10 | 3 | 13
  Race: White | 439 | 450 | 889
  Race: Not reported | 7 | 9 | 16
  Race: Other | 5 | 8 | 13
Weight [Mean (Standard Deviation); unit: kg] — Population: Not all subject in the safety population had valid weights collected at Baseline
  kg
    number analyzed (Participants) | 465 | 471 | 936
    (all) | 77.76 (16.008) | 77.21 (15.027) | 77.48 (15.516)
Height [Mean (Standard Deviation); unit: cm] | 172.0 (10.22) | 172.0 (9.30) | 172.0 (9.77)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: Not all subject in the safety population had valid weights collected at Baseline, therefore BMI could not be calculated.
  kg/m^2
    number analyzed (Participants) | 465 | 471 | 936
    (all) | 26.15 (4.330) | 26.00 (4.239) | 26.08 (4.283)
ALS family history [Count of Participants; unit: Participants]
  Yes | 26 | 33 | 59
  No | 442 | 440 | 882
  Missing | 0 | 1 | 1
Time since ALS symptom onset [Mean (Standard Deviation); unit: months] | 15.53 (5.411) | 14.92 (5.251) | 15.22 (5.337)
Site of onset [Count of Participants; unit: Participants]
  Bulbar | 112 | 107 | 219
  Other | 356 | 367 | 723
Time since ALS diagnosis [Mean (Standard Deviation); unit: months] | 7.62 (5.015) | 7.22 (4.718) | 7.42 (4.869)
El Escorial Criteria for ALS [Count of Participants; unit: Participants]
  Possible | 44 | 44 | 88
  Probable laboratory supported | 94 | 98 | 192
  Probable | 174 | 185 | 359
  Definite | 156 | 147 | 303
Concomitant use of riluzole [Count of Participants; unit: Participants]
  Yes | 349 | 359 | 708
  No | 119 | 115 | 234
Baseline ALSFRS-R total scores [Mean (Standard Deviation); unit: units on a scale] — Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R). This validated scale stratifies severity of amyotrophic lateral sclerosis (ALS). The ALSFRS-R consists of 12 items answered across 4 functional domains (bulbar, gross motor, fine motor and respiratory) in which each item is scored between 4 and 0, for a maximum score of 48. A decline in ALSFRS-R indicates a loss of physical function.
  units on a scale | 37.9 (5.65) | 38.4 (5.24) | 38.2 (5.45)
Baseline predicted upright slow vital capacity (%) [Count of Participants; unit: Participants] — slow vital capacity
  Participants
    <65% | 27 | 28 | 55
    65-75% | 84 | 79 | 163
    >75% | 357 | 367 | 724
Baseline predicted upright slow vital capacity (%) [Mean (Standard Deviation); unit: %] — slow vital capacity
  % | 89.1 (17.71) | 89.0 (17.57) | 89.1 (17.63)

OUTCOME MEASURES:

1. Primary Outcome: Composite Assessment of Function and Survival (CAFS) at 12 Months
Description: The Composite Assessment of Function and Survival (CAFS) is a between-group comparison of a single ranked clinical outcome based on (1) the change from baseline in ALS Functional Rating Scale-Revised (ALSFRS-R) score and (2) time to death. Each subject is ranked according to time-to-death (earlier deaths ranked lower than later deaths). Subjects who survive are ranked more favorably than subjects who died. Among the survivors, subjects are ranked according to change in ALSFRS-R (greater worsening of ALSFRS-R is ranked lower than less worsening or an improvement in ALSFRS-R). The ranked scores range from 001 to 941 (the number of subjects in the Efficacy Population) with larger rank score numbers associated with a better outcome. The ranks were analyzed using an ANCOVA model, which includes treatment as a fixed effect and adjusts for baseline ALSFRS-R score, duration of symptoms, site of onset, and use of riluzole. The least square mean rank score is presented for each treatment group.
Time Frame: 12 months
Population: The efficacy population is defined as subjects who were randomized and received at least 1 dose of study treatment and who either had at least 1 available post-dosing efficacy evaluation (ALSFRS-R) or died during the study period. Subjects were analyzed in the treatment group to which they are randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dexpramipexole
Number analyzed (Participants) | 468 | 473
units on a scale | 438.84 [412.807 to 464.878] | 441.76 [415.426 to 468.084]
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole; Test type: Superiority; p = 0.8568, ANCOVA; Includes treatment as a fixed effect and adjusts for baseline ALSFRS-R total score, duration from sx onset, site of onset, and use of riluzole; LS Mean Difference (Final Values) = 2.91, 95% CI 2-sided [-28.751 to 34.576]

2. Primary Outcome: Death up to 12 Months (CAFs Individual Component)
Description: The longest duration of follow-up for this time to the death analysis was 12 months. In the study, subjects were followed for 12-18 months.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dexpramipexole
Number analyzed (Participants) | 468 | 473
percentage of participants | 17.2 | 16.0
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole; Test type: Superiority; p = 0.8375, Cox Proportional Hazards model; Adjusted for baseline ALSFRS-R total score, duration from symptom onset to the first dose of study treatment, site of onset, and use of riluzole; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.750 to 1.427]; Hazard Ratio (HR) (Dex/PBO)

3. Primary Outcome: Change From Baseline in ALSFRS-R at 12 Months (CAFs Individual Component)
Description: The ALSFRS-R (ALS functional rating scale with respiratory component) is a validated scale which measures 4 functional domains, comprising respiratory function, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score of 48, with higher scores representing better function.
Time Frame: 12 months
Population: The efficacy population is defined as subjects who were randomized and received at least 1 dose of study treatment and who either had at least 1 available post-dosing efficacy evaluation (ALSFRS-R) or died during the study period. Subjects will be analyzed in the treatment group to which they are randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dexpramipexole
Number analyzed (Participants) | 468 | 473
units on a scale | -13.415 [-14.275 to -12.555] | -13.339 [-14.199 to -12.480]
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole; Test type: Superiority; p = 0.9019, mixed-effects repeated-measures model; Mixed-effects repeated-measures model with treatment, visit, treatment-by visit interaction, baseline ALSFRS-R score, baseline-by-visit interaction; LS Mean Difference (Net) = 0.076, 95% CI 2-sided [-1.128 to 1.280] — The mixed-effects repeated-measures model also adjusted for the following covariates: duration from symptom onset, site of onset, and use of riluzole

4. Secondary Outcome: Death or Respiratory Insufficiency (DRI) up to Month 18
Description: Time to Death or Respiratory Insufficiency (DRI) is defined as receipt of a tracheostomy or the use of non-invasive ventilation (NIV) for ≥22 hours per day for at least 10 consecutive days. If NIV is used to meet the criteria for respiratory insufficiency, no measured slow vital capacity (SVC) at any subsequent assessment may be >50%. Time to DRI is calculated from the date of the first dose to the first date of one of the following events: death, tracheostomy, or the 10th day of consecutive NIV with no measured SVC >50% at any subsequent assessment.
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dexpramipexole
Number analyzed (Participants) | 468 | 474
percentage of participants | 27.2 | 22.3
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole; Test type: Superiority; p = 0.7715, Cox Proportional Hazards model; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.801 to 1.348]

5. Secondary Outcome: Death up to 18 Months
Description: Estimated time to death up to 18 months. This includes deaths reported greater than 30 days following discontinuation from the study (the time period for reporting all-cause mortality), regardless of subject disposition, up to 18 months from first dose.
Time Frame: 18 months
Population: Subjects who were randomized, received at least 1 dose of study treatment, had at least 1 available post-dosing efficacy evaluation (ALSFRS-R) or died during the study period. Subjects were analyzed in the treatment group to which they are randomized. An attempt was made to collect living status for each subject 18 months after randomization, regardless of the subject's disposition in the study (active or discontinued) or primary reasons for discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dexpramipexole
Number analyzed (Participants) | 468 | 474
percentage of participants | 23.1 | 20.5
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole; Test type: Superiority; p = 0.9033, Cox Proportional Hazards model; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.745 to 1.298]

6. Secondary Outcome: ≤50% Predicted Upright Slow Vital Capacity (SVC) or Died up to 18 Months
Description: The date of reaching ≤50% of predicted upright slow vital capacity (SVC) is defined as the date of the first visit at which a predicted upright SVC is ≤50% and continues to remain ≤50% at the subsequent visit except for the last available observation. The time to reach ≤50% of predicted upright SVC is defined as the duration between the date of reaching ≤50% of predicted upright SVC and the date of the first dose of study medication. If the subject is alive and does not reach ≤50% of predicted upright SVC, the time to reach ≤50% of predicted upright SVC will be censored and equal to the number of days from the first dose of study medication until the visit date when the subject's last available SVC assessment is performed. The earliest time (Reaching ≤50% Predicted Upright SVC or death) is used in analysis.
Time Frame: 18 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dexpramipexole
Number analyzed (Participants) | 468 | 474
percentage of participants | 41.9 | 36.5
Statistical Analysis 1: Comparison: Placebo vs Dexpramipexole; Test type: Superiority; p = 0.7720, Cox Proportional Hazards model; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.789 to 1.192] — Hazard ratio (Dex/PBO)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Placebo | Dexpramipexole
All-Cause Mortality (participants affected / at risk) | 108/468 | 97/474
Serious Adverse Events (participants affected / at risk) | 233/468 | 225/474
Other Adverse Events (participants affected / at risk) | 447/468 | 459/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=468) | Dexpramipexole (N=474)
PNEUMONIA (Infections and infestations) | 19 | 14
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 3
URINARY TRACT INFECTION (Infections and infestations) | 3 | 3
BRONCHITIS (Infections and infestations) | 6 | 2
CELLULITIS (Infections and infestations) | 0 | 2
LUNG INFECTION (Infections and infestations) | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2
CATHETER SITE INFECTION (Infections and infestations) | 1 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 1
CYSTITIS ESCHERICHIA (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
NEUTROPENIC INFECTION (Infections and infestations) | 0 | 1
PILONIDAL CYST (Infections and infestations) | 0 | 1
PSEUDOMONAS BRONCHITIS (Infections and infestations) | 0 | 1
RHINITIS (Infections and infestations) | 0 | 1
RHINOVIRUS INFECTION (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
GAS GANGRENE (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
PNEUMONIA KLEBSIELLA (Infections and infestations) | 2 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS BRONCHITIS (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
SEPSIS (Infections and infestations) | 1 | 0
SERRATIA INFECTION (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 9
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 2
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 1
ALCOHOLISM (Psychiatric disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 | 0
PANIC ATTACK (Psychiatric disorders) | 1 | 0
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 16 | 16
MOTOR NEURONE DISEASE (Nervous system disorders) | 7 | 3
MIGRAINE (Nervous system disorders) | 0 | 1
MUSCLE SPASTICITY (Nervous system disorders) | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 2 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
BULBAR PALSY (Nervous system disorders) | 1 | 0
CEREBELLAR INFARCTION (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
VERTEBRAL ARTERY DISSECTION (Nervous system disorders) | 1 | 0
CATARACT (Eye disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 3 | 5
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 4
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 3
ARRHYTHMIA (Cardiac disorders) | 0 | 2
CARDIAC ARREST (Cardiac disorders) | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 0 | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 1
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 2 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 8 | 8
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 75 | 69
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 13 | 12
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 9 | 12
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 | 6
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 5 | 4
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 6 | 4
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 6 | 3
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 6 | 2
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH DECREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 4 | 1
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INCREASED BRONCHIAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 3 | 1
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY MUSCLE WEAKNESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INCREASED VISCOSITY OF BRONCHIAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VOCAL CORD DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 69 | 62
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2
APHAGIA (Gastrointestinal disorders) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 4 | 2
FAECALOMA (Gastrointestinal disorders) | 0 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 2 | 0
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 | 1
INCLUSION BODY MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
NOSE DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 3
URINARY RETENTION (Renal and urinary disorders) | 1 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
URETERIC STENOSIS (Renal and urinary disorders) | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 1
BREAST HAEMATOMA (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
EUTHANASIA (General disorders) | 1 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 2
SUDDEN DEATH (General disorders) | 0 | 2
ADVERSE DRUG REACTION (General disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 1
CATHETER SITE HAEMORRHAGE (General disorders) | 0 | 1
CHEST PAIN (General disorders) | 0 | 1
COMPLICATION OF DEVICE INSERTION (General disorders) | 0 | 1
DEATH (General disorders) | 1 | 1
DEVICE MALFUNCTION (General disorders) | 0 | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 1
ULCER HAEMORRHAGE (General disorders) | 0 | 1
DEVICE LEAKAGE (General disorders) | 1 | 0
DEVICE OCCLUSION (General disorders) | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
VITAL CAPACITY DECREASED (Investigations) | 3 | 3
WEIGHT DECREASED (Investigations) | 1 | 2
INVESTIGATION (Investigations) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1
DIAGNOSTIC PROCEDURE (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0
OXYGEN SATURATION DECREASED (Investigations) | 2 | 0
TOTAL LUNG CAPACITY DECREASED (Investigations) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 11 | 13
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
LACERATION (Injury, poisoning and procedural complications) | 1 | 2
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 3 | 2
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 2 | 1
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPLENIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1 | 0
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 2 | 0
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
TRENCH FOOT (Injury, poisoning and procedural complications) | 1 | 0
SUPPORTIVE CARE (Surgical and medical procedures) | 1 | 0
RESPITE CARE (Social circumstances) | 1 | 0
SOCIAL STAY HOSPITALISATION (Social circumstances) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=468) | Dexpramipexole (N=474)
NASOPHARYNGITIS (Infections and infestations) | 76 | 69
URINARY TRACT INFECTION (Infections and infestations) | 56 | 56
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 | 30
PNEUMONIA (Infections and infestations) | 32 | 24
BRONCHITIS (Infections and infestations) | 28 | 21
NEUTROPENIA (Blood and lymphatic system disorders) | 8 | 37
DECREASED APPETITE (Metabolism and nutrition disorders) | 27 | 33
INSOMNIA (Psychiatric disorders) | 60 | 71
DEPRESSION (Psychiatric disorders) | 50 | 40
ANXIETY (Psychiatric disorders) | 34 | 35
HEADACHE (Nervous system disorders) | 65 | 66
DIZZINESS (Nervous system disorders) | 28 | 42
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 28 | 24
HYPERTENSION (Vascular disorders) | 13 | 23
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 81 | 72
COUGH (Respiratory, thoracic and mediastinal disorders) | 30 | 45
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 52 | 44
CONSTIPATION (Gastrointestinal disorders) | 109 | 129
NAUSEA (Gastrointestinal disorders) | 65 | 106
DYSPHAGIA (Gastrointestinal disorders) | 95 | 88
DIARRHOEA (Gastrointestinal disorders) | 55 | 44
DRY MOUTH (Gastrointestinal disorders) | 20 | 41
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 34 | 29
RASH (Skin and subcutaneous tissue disorders) | 27 | 27
PRURITUS (Skin and subcutaneous tissue disorders) | 18 | 25
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 44 | 64
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 37 | 44
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 34 | 42
BACK PAIN (Musculoskeletal and connective tissue disorders) | 36 | 39
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 30 | 38
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 28 | 26
NECK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 24
OEDEMA PERIPHERAL (General disorders) | 72 | 61
FATIGUE (General disorders) | 60 | 57
ASTHENIA (General disorders) | 10 | 23
PYREXIA (General disorders) | 21 | 22
WEIGHT DECREASED (Investigations) | 48 | 75
FALL (Injury, poisoning and procedural complications) | 198 | 192
LACERATION (Injury, poisoning and procedural complications) | 31 | 34
CONTUSION (Injury, poisoning and procedural complications) | 35 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must be consulted